CLINICAL TRIAL: NCT05140655
Title: Real-world Effectiveness and Safety of a Generic Fulvestrant Alone or in Combination With Cyclin Inhibitors in Postmenopausal Women With Advanced Breast Cancer HR+, HER2-, in Two Colombian Referral Centers
Brief Title: Effectiveness and Safety of Fulvestrant in Postmenopausal Women With Advanced Breast Cancer HR+, HER2-
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Reddy's Laboratories SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: DRLCOLCT001
Record Dates: First submitted 2021-11-11; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Breast Neoplasm Female
MeSH Terms: interventions — Fulvestrant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Fulvestrant — Medicine for Advanced breast cancer

SUMMARY:
A phase IV, single arm study will be performed in postmenopausal women with locally advanced or metastatic breast cancer. All patients included will receive fulvestrant from Dr. Reddy's Laboratories, in accordance with local practice and the regulatory authorization of the drug in Colombia. This study will be carried out for 1 year and approximately 40 patients will be included in 2 research centers selected for its conduct.

Patients who meet the inclusion criteria and who do not have to be discarded from entering the study due to meeting any of the exclusion criteria, will be evaluated to determine the effectiveness and tolerability of the administration of Dr. Reddy's fulvestrant at a dose of 500 mg / month plus an additional indicated dose 14 days after the initial dose, for 12 months of follow-up or until disease progression or the appearance of unacceptable toxicity. The assessment of tolerability will be carried out based on the collection of data related to adverse events from the first dose administered.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women (defined as those with permanent cessation of menstruation for more than 12 months, regardless of whether their menopausal condition occurred naturally or was artificially induced), ambulatory or hospitalized
2. Diagnosis of advanced breast cancer HR +, HER2-
3. Positivity for hormone receptors (either estrogen, progesterone, or both).
4. Negative for human epidermal growth factor receptor 2 (HER2).
5. Acceptance of informed consent, if it is required by local regulatory standards.

Exclusion Criteria

1. History of previous treatment with fulvestrant.
2. Concomitant treatment with antitumor drugs other than cyclin inhibitors (abemaciclib, palbociclib, ribociclib).
3. Pregnancy.
4. Lactation.
5. Hypersensitivity to any of the excipients included in the complete formulation of fulvestrant from Dr. Reddy's Laboratories Limited.
6. Renal insufficiency grade 4 or 5 (creatinine clearance <30 ml / min / 1.73 m2 according to the classification of the National Kidney Foundation).
7. Hepatic failure (Child-Pugh C stage).
8. Performance status ECOG ≥ 3.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal Women with Advanced Breast Cancer HR+, HER2-
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-04-19 (Estimated); Study Completion 2022-08-19 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Measured at 12 months
  Objective response rate (ORR), defined as the proportion of patients with a complete response or partial response to treatment according to Response Evaluation Criteria in Solid Tumors (RECIST)percentage of patients with complete response or partial response) according to RECIST 1.1
Clinical benefit rate (percentage of patients with complete response, partial response and stable disease) | Measured at 12 months
  CBR is the proportion of patients with a complete or partial response or with stable disease
Overall survival rate | 12 months
  The percentage of people in a study or treatment group who are still alive for a certain period of time after they were diagnosed with or started treatment for a disease
Disease-free survival rate | 12 months
  It is the percentage of individuals in the treatment group who are likely to be free of the signs and symptoms of a disease after a specified duration of time

SECONDARY OUTCOMES:
Describe the demographic characteristics of the patients included in the study | Measured at 12 months
Assess percentage of patients with adverse events (assessed by CTCAEv4.0) from the first administration and until the end of follow-up. | Measured at 12 months
  Common Terminology Criteria for Adverse Events
Assess Percentage of patients with serious adverse events (assessed by CTCAEv4.0) from the first administration to the end of follow-up. | Measured at 12 months
  Common Terminology Criteria for Adverse Events
Assess incidence, severity, and relationship to treatment defined by the investigator for reported adverse events. | Measured at 12 months
  Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Ray Manneh, Principal Investigator — SOHEC; José Lobatón, Principal Investigator — IMAT
Locations (1):
- SOHEC, Valledupar, Cesar Department, Colombia

IPD SHARING:
Plan to Share IPD: No